CLINICAL TRIAL: NCT00348933
Title: Efficacy of a Therapeutic Treatment Trial in Angelman Syndrome
Brief Title: Dietary Supplements for the Treatment of Angelman Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Baylor College of Medicine (Other); Rady Children's Hospital, San Diego (Other); Boston Children's Hospital (Other); Greenwood Genetic Center (Other); Rare Diseases Clinical Research Network (Network)
Responsible Party: Principal Investigator, Lynne M. Bird, Principal Investigator, University of California, San Diego
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDCRN 5204
Record Dates: First submitted 2006-07-03; First posted 2006-07-06 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Angelman Syndrome; Nervous System Diseases
Keywords: Developmental Delay; Mental Retardation; Ataxia; Microcephaly; Seizures
MeSH Terms: conditions — Angelman Syndrome; Nervous System Diseases; Learning Disabilities; Intellectual Disability; Ataxia; Microcephaly; Seizures | interventions — Betaine; Creatine; levomefolate calcium; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive two daily doses of Metafolin, betaine, and creatine, and one daily dose of vitamin B12 for 12 months.
  Interventions: Drug: Betaine; Drug: Creatine; Drug: Metafolin; Drug: Vitamin B12

INTERVENTIONS:
Drug: Betaine — 100-200 mg per kg per day by mouth with a maximum of 6 grams divided in two daily doses
Drug: Creatine — 200 mg per kg per day with a daily maximum of 5 grams divided in two daily doses
Drug: Metafolin — 0.5 mg per kg per day by mouth with a maximum of 8 milligrams divided in two daily doses
Drug: Vitamin B12 — 1 mg by mouth per day for all weights and ages

SUMMARY:
Angelman syndrome (AS) is a complex genetic disorder that affects the nervous system. The purpose of this study is to determine the effectiveness of certain dietary supplements in treating the symptoms of AS.

DETAILED DESCRIPTION:
AS is a neurologic disorder that may cause developmental delay, mental retardation, severe speech impairment, seizures, small head size, and problems with movement and balance in young children. AS is caused by a missing or incomplete chromosome 15 that is inherited from the mother. Diagnosis of AS is usually made between three and seven years of age, when the characteristic behaviors and features of the disease become most evident. Prior to AS diagnosis, the symptoms may be mistaken for cerebral palsy or autism. Physical, occupational, and speech therapy, communication skills development, and behavior modification help to improve the quality of life of these children, but other treatments are needed.

In a previous study, decreased DNA methylation, which is a type of chemical change in DNA, was observed in an individual with AS; this condition may be a primary cause of AS. It is hypothesized that promoting increased DNA methylation might reduce the severity of AS symptoms. Betaine, creatine, Metafolin, and vitamin B12 are compounds normally found in the body that are involved in the DNA methylation pathway. Increasing the concentrations of these compounds in the body may enhance DNA methylation. This study will evaluate the efficacy of four dietary supplements in treating the symptoms of AS.

This study will last 12 months. Study visits will occur at study entry and Month 12. A selected group of participants, those who meet the diagnostic criteria for autism, will also be evaluated at Month 6. At study visits, participants will undergo an electroencephalogram (EEG). Medical history, physical exam, neurological exams, and developmental assessments will also be performed. Urine and blood collection, including tests to determine the blood levels of the dietary supplements, will occur at study entry and Months 6 and 12. Participants will receive two daily doses of Metafolin, betaine, and creatine, and one daily dose of vitamin B12 for the duration of the study. Parents will be asked to complete a questionnaire at each visit to report their child's behavior while taking the dietary supplements. Parents will also be contacted by phone periodically to assess changes and/or progress in their children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AS
* In stable condition with relatively good control of seizures
* Willing to comply with treatment, study visit schedule, and study assessments
* Willing to take oral or G-tube medication
* Willing to be contacted monthly during the course of the study
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* History of liver or kidney disease
* Currently being treated for a serious acute illness
* Known hypersensitivity to any of the study drugs
* Received high-dose folate drug treatment in the 12 months prior to study entry
* Other significant medical problems, including those involving the liver, kidney, or heart
* Other comorbidities, genetic disorders, or extreme prematurity; children with autism are not excluded

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2006-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L. Beaudet, MD, Principal Investigator — Department of Molecular and Human Genetics, Baylor College of Medicine; Carlos A. Bacino, MD, Principal Investigator — Department of Molecular and Human Genetics, Baylor College of Medicine; Wen-Hann Tan, BMBS, Principal Investigator — Harvard Medical School, Children's Hospital Boston; Lynne M. Bird, MD, Principal Investigator — Division of Dysmorphology/Genetics, Children's Hospital San Diego, Department of Pediatrics, University of California, San Diego; Steven A. Skinner, MD, Principal Investigator — Greenwood Genetic Center
Locations (4):
- United States (4):
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Greenwood Genetics Center, Greenwood, South Carolina
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Kishino T, Lalande M, Wagstaff J. UBE3A/E6-AP mutations cause Angelman syndrome. Nat Genet. 1997 Jan;15(1):70-3. doi: 10.1038/ng0197-70. PMID 8988171
- [Background] Williams CA, Beaudet AL, Clayton-Smith J, Knoll JH, Kyllerman M, Laan LA, Magenis RE, Moncla A, Schinzel AA, Summers JA, Wagstaff J. Angelman syndrome 2005: updated consensus for diagnostic criteria. Am J Med Genet A. 2006 Mar 1;140(5):413-8. doi: 10.1002/ajmg.a.31074. PMID 16470747
- [Background] Williams CA, Lossie A, Driscoll D; R.C. Phillips Unit. Angelman syndrome: mimicking conditions and phenotypes. Am J Med Genet. 2001 Jun 1;101(1):59-64. doi: 10.1002/ajmg.1316. PMID 11343340
- [Derived] Han J, Bichell TJ, Golden S, Anselm I, Waisbren S, Bacino CA, Peters SU, Bird LM, Kimonis V. A placebo-controlled trial of folic acid and betaine in identical twins with Angelman syndrome. Orphanet J Rare Dis. 2019 Oct 22;14(1):232. doi: 10.1186/s13023-019-1216-0. PMID 31640736
- [Derived] Bird LM, Tan WH, Bacino CA, Peters SU, Skinner SA, Anselm I, Barbieri-Welge R, Bauer-Carlin A, Gentile JK, Glaze DG, Horowitz LT, Mohan KN, Nespeca MP, Sahoo T, Sarco D, Waisbren SE, Beaudet AL. A therapeutic trial of pro-methylation dietary supplements in Angelman syndrome. Am J Med Genet A. 2011 Dec;155A(12):2956-63. doi: 10.1002/ajmg.a.34297. Epub 2011 Oct 14. PMID 22002941

RESULTS

PARTICIPANT FLOW:
Groups:
- Metafolin, Betaine, Creatine, B12 Treatment: Participants will receive two daily doses of Metafolin, betaine, and creatine, and one daily dose of vitamin B12 for 12 months.
Period: Overall Study
Arm/Group | Metafolin, Betaine, Creatine, B12 Treatment
Started | 90
Completed | 65
Not Completed | 25
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Metafolin, Betaine, Creatine, B12 Treatment
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 90
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 2.9 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Functioning in Specific Areas of Development, Including Speech and Communications Skills, Cognitive Abilities and Daily Living Skills
Description: Primary:
  Bayley Scales of Infant Development measures Mental Developmental Index standard scores 0 (least skilled) - 100 (most skilled) Psychomotor Developmental Index standard scores 0 (least skilled - 10 (most skilled) Vineland Adaptive Behavior Scales (VABS), Communication standard scores 0 (least skilled) - 100 (most skilled) Daily Living Skills standard scores 0 (least skilled) - 100 (most skilled) Socialization standard scores 0 (least skilled) - 100 (most skilled) Motor Skills standard scores 0 (least skilled) - 100 (most skilled) Preschool Language Scale (PLS), Auditory Comprehension 0 (least skilled) - 100 (most skilled) Expressive Communication 0 (least skilled) - 100 (most skilled)
Time Frame: Baseline, 1 year
Population: Analysis per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment (Metafolin/Creatine/Betaine/B12)
Number analyzed (Participants) | 65
units on a scale
  Bayley Scales Mental Developmental Index | 5.7 (7.8)
  Bayley Scales Psychomotor Developmental Index | 4.7 (8.6)
  VABS Communication | 5.8 (8.3)
  VABS Daily Living Skills | 3.7 (7.9)
  VABS Socialization | 4.7 (5.2)
  VABS Motor Skills | 2.0 (6.1)
  PLS Auditory Comprehension | 2.0 (10.8)
  PLS Expressive Communication | 5.5 (9.6)

2. Secondary Outcome: Change in Levels of Betaine, Creatine, Dimethylglycine, Guanidinoacetate, Homocysteine, and Methionine.
Time Frame: Baseline, 1 year
Population: analysis per protocol
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Treatment (Metafolin/Creatine/Betain/B12): All participants received treatment. Compared to a placebo group from a previous study.
Arm/Group | Treatment (Metafolin/Creatine/Betain/B12)
Number analyzed (Participants) | 65
mmol/L
  Betaine | 206.9 (224.5)
  Creatine | 83.3 (165.9)
  Dimethylglycine | 93.7 (129)
  Guanidinoacetate | 0.11 (0.34)
  Homocysteine | 2.3 (2.1)
  Methionine | 5.5 (12.1)

3. Secondary Outcome: Change in RBC Folate
Time Frame: Baseline, 1 year
Population: Analysis per protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (Metafolin/Creatine/Betaine/B12)
Number analyzed (Participants) | 65
ng/mL | 77 (267)

ADVERSE EVENTS:
Arm/Group | Metafolin, Betaine, Creatine, B12 Treatment
Serious Adverse Events (participants affected / at risk) | 48/90
Other Adverse Events (participants affected / at risk) | 5/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metafolin, Betaine, Creatine, B12 Treatment (N=90)
Seizure (Nervous system disorders) | 18 (18)
Insomnia (General disorders) | 14 (14)
Constipation (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Behavior disturbance (Psychiatric disorders) | 2 (2)
Infection (Infections and infestations) | 7 (7)
Serum sickness (Immune system disorders) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metafolin, Betaine, Creatine, B12 Treatment (N=90)
Laboratory abnormalities (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Body Odor (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No